CLINICAL TRIAL: NCT04543045
Title: Qualitative Exploration of Head & Neck Cancer Patient Reported Experience of Radiotherapy With Focus on Restriction Anxiety & 'Claustrophobia
Brief Title: Qualitative Exploration of Head & Neck Cancer Patient Reported Experience of Radiotherapy
Acronym: H&NPRER-RAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp182
Record Dates: First submitted 2020-07-30; First posted 2020-09-09 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Oncology; Head and Neck Cancer; Anxiety
Keywords: patient experience; claustrophobia; radiotherapy; radiotherapy moulds; radiotherapy masks
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Anxiety Disorders; Claustrophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: 20 patients will be interviewed once, which will be approximately 60 minutes in duration. The interviews will be audio recorded.
  Interventions: Other: not an intervention
- Stage 2: Five patients who participated in stage 1 will take part in a cognitive interview, which will be approximately 60 minutes in duration.The interviews will be audio recorded.
  Interventions: Other: not an intervention

INTERVENTIONS:
Other: not an intervention — not an intervention

SUMMARY:
The study aims to explore the experience of patients with Head and Neck Cancer, who are preparing for and/or completed radiotherapy treatment.

DETAILED DESCRIPTION:
This is a non-interventional study using interviews to explore head and neck cancer patients' experience of preparing for and completing radiotherapy utilising an immobilisation mask.

The study will be conducted in 2 stages:

The first stage is Item generation. Approximately 20 interviews will be conducted with head and neck cancer patients who have completed or partially completed radiotherapy. The interviews will capture their experiences and views pertaining to mould making, scans and radiotherapy, reported associated fear of restriction, suffocation, loss of control and fear of public embarrassment during treatment.

The data from the interviews will be used to develop potential items for a screening tool for identification of those patients likely to experience anxiety and claustrophobia before they start their treatment.

The second stage is cognitive interviews. Approximately 5 patients included in Stage I will be invited to take part in a further interview to review the themes and potential questionnaire items identified from interviews.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 (no upper age limit)
* Completed or partially completed radiotherapy treatment utilising a mask ≥ 6 weeks previous to study entry

Exclusion Criteria:

* Unable to understand and communicate in the English language
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Range of patients who have completed or partially completed radiotherapy treatment utilising a mask. This will include a range of patients (i) those who's records indicate, or patients report that they experienced severe difficulties tolerating the mask, (ii) those who could not complete the full course of radiotherapy; and (iii) those who experienced no difficulties at all.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Patient experience | within 6 weeks of using a mask
  Interviews will be used to generate themes that capture the patients experience. These themes are the primary outcome.There are no units of measurement or data collection tools only an interview schedule.

SECONDARY OUTCOMES:
potential items for a questionnaire | 2 months after completing or partially completing radiotherapy.
  interviews extracts will be used as potential item for the interview

CONTACTS AND LOCATIONS:
Overall Officials: Jacqui Stringer, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No